CLINICAL TRIAL: NCT01220804
Title: Evaluation of Blood-retinal Barrier Functional Alterations by Optical Coherence Tomography
Acronym: CNTM025A OCT
Status: Completed | Type: Observational
Sponsor: Association for Innovation and Biomedical Research on Light and Image (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other); Instituto Financeiro para o Desenvolvimento Regional (Unknown)
Responsible Party: Sponsor
Other Study IDs: PTDC/SAU-BEB/103151/2008
Record Dates: First submitted 2010-10-11; First posted 2010-10-14 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- NPDR: Type 2 diabetic patients with nonproliferative diabetic retinopathy (NPDR)
- Control Population: Healthy volunteers

SUMMARY:
The purpose of this study is to identify alterations of the blood-retinal barrier (BRB) in diabetic retinas using a novel non-invasive approach based on the Fourier domain high-definition optical coherence tomograph (OCT).

DETAILED DESCRIPTION:
Type 2 diabetic patients with nonproliferative diabetic retinopathy (NPDR) (study population) and healthy volunteers (control population).

Inclusion Criteria:

Age over 18 years; type-2 diabetes; NPDR levels 10, 20 and 35/47 (ETDRS severity scale); and an area of retinal leakage of at least 25% of the RLA map (macular area).

Exclusion Criteria:

Presence of media opacity; vitreous syneresis or posterior vitreous detachment, and; previous photocoagulation treatments or any type of intraocular surgery or intravitreal medications; and other retinal pathologies.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years; type-2 diabetes; NPDR levels 10, 20 and 35/47 (ETDRS severity scale), and area of retinal leakage of at least 25% of the RLA map (macular area).

Exclusion Criteria:

* Presence of media opacity; vitreous syneresis or posterior vitreous detachment, and; previous photocoagulation treatments or any type of intraocular surgery or intravitreal medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Type 2 diabetic patients with nonproliferative diabetic retinopathy (NPDR) (study population) and healthy volunteers (control population).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2010-11; Primary Completion 2011-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Optical reflectivity as measured by optical coherence tomography | 14 months
  To analyse OCT reflectivity distribution between areas with and without fluorescein leakage in type 2 diabetic eyes. In previous studies our group found differences, when comparing the histograms of the optical reflectivity distribution, suggesting that the optical reflectivity, as measured by OCT, may change under BRB alterations

CONTACTS AND LOCATIONS:
Locations (1):
- AIBILI, Coimbra, Portugal

REFERENCES:
- See also: Related Info — http://www.aibili.pt